CLINICAL TRIAL: NCT04452461
Title: MFOLFIRINOX or Gemcitabine / Nab-paclitaxel Followed by Pancreatectomy for Patients with Borderline Resectable Pancreatic Adenocarcinoma. a Pilot Feasibility Study.
Brief Title: Pancreatic Adenocarcinoma Neoadjuvant Chemotherapy Before Surgery
Acronym: PANCREAS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Pablo Serrano, Associate Professor, Hamilton Health Sciences Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5076
Record Dates: First submitted 2020-06-22; First posted 2020-06-30 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Pancreatic Adenocarcinoma
MeSH Terms: interventions — Fluorouracil; Leucovorin; Oxaliplatin; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm Intervention (Other): 1. Chemotherapy: 6 cycles (three months) of IV combination chemotherapy with mFOLFIRINOX on day 1 followed by one week of rest (14-day cycle). Alternatively, patients will receive three months of gemcitabine / nab-paclitaxel.
  2. Re-staging CT scan with Carbohydrate Antigen (CA) 19-9 serum test.
  3. Staging laparoscopy to rule out occult metastatic disease is optional based on surgeon's preference.
  5. Pancreatectomy 4 weeks following the last day of Chemotherapy as per standard of care.
  6. Adjuvant chemotherapy: as per standard of care. 7. Clinical assessment and CT scan with CA 19-9 serum test at 4-month intervals until identification of cancer recurrence.
  8. Follow up of patients after 2 years every six months for up to 5 years following the initiation of treatment will be performed off-protocol as per standard of care.
  Interventions: Drug: mFOLFIRINOX; Drug: Gemcitabine / Nab-paclitaxel

INTERVENTIONS:
Drug: mFOLFIRINOX — mFOLFIRINOX, including: Oxaliplatin 85 mg/m2 IV over 2 hours, Leucovorin 400mg/m2 IV over 2 hours, Irinotecan at 150 mg/m2 IV over 90 min, 5-Fluoruracil continuous infusion of 2400 mg/m2 IV over 46h.
  Other Names: 5-FU; leucovorin; oxaliplatin
Drug: Gemcitabine / Nab-paclitaxel — Both drugs are administered once weekly for three weeks (days 1, 8, 15) followed by a week of rest (28-day cycle) for 3 cycles prior to imaging. Gemcitabine: 1000 mg/m2 intravenous infusion over 30 to 40 minutes. Nab-paclitaxel: 125 mg/m2 intravenous infusion over 30 to 40 minutes.
  Other Names: gemcitabine / abraxane

SUMMARY:
This is a single-arm, single-center feasibility trial of patients with borderline resectable pancreatic adenocarcinoma receiving chemotherapy with mFOLFIRINOX or gemcitabine / nab-paclitaxel followed by pancreatectomy.

DETAILED DESCRIPTION:
Borderline resectable pancreatic adenocarcinoma infiltrates into adjacent vascular structures to an extent such that complete macroscopic resection is technically feasible, but an R0 resection poses a challenge when surgery is the primary therapy. Therefore, a different management strategy may be beneficial.

The primary outcome of the PANCREAS trial is defined as the proportion of eligible patients enrolled in the study over an 18-month period and the proportion of patients who complete the protocol (neoadjuvant therapy and pancreatectomy). Certain modifications of the neoadjuvant therapy protocol are expected and allowed, and the primary feasibility outcome will be one of the following: stop, main study non-feasible; continue with protocol modifications; or continue without modification. A safety analysis will be performed after first 15 patients are enrolled and complete neoadjuvant therapy and surgery. Patients enrolled in this trial will undergo interventions in the following order: neoadjuvant chemotherapy, re-staging CT scan, pancreatectomy and adjuvant chemotherapy. Postoperative mortality will be recorded up to 90 days after surgery. Patients will be followed every four months with a CT scan of the chest/abdomen for two years after resection or until evidence of disease recurrence. Patients who do not undergo surgical resection will be followed for two years after accrual (duration of study period) or until evidence of disease progression or death.

ELIGIBILITY:
Inclusion Criteria:

* 1. Men and women 18 years of age or older who present with biopsy proven borderline resectable pancreatic adenocarcinoma who are medically fit for surgery as per assessment by treating surgeon.

  2. Age ≤ 79 years 3. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 4. Normal bone marrow and organ function
  1. Absolute neutrophil count (ANC) = or > 1500, platelets > 100K
  2. Total bilirubin <1.5x upper limit of normal (ULN)
  3. Alanine transaminase (ALT), Aspartate aminotransferase (AST) < 3 x ULN
  4. Creatinine <150umol/L
  5. Normal prothrombin time and international normalized ratio (INR) 5. Able to provide written informed consent

Exclusion Criteria:

1. Proven metastatic disease (e.g. on imaging modality such as CT scan of the chest, abdomen and pelvis or MRI)
2. Locally advanced pancreatic cancer (see definition section 3.3)
3. Prior treatment with radiation therapy to the pancreas or associated field.
4. Contraindications to receive chemotherapy
5. History of cardiac disease including congestive heart failure (New York Heart Association class 2), active coronary artery disease or uncontrolled hypertension
6. Concurrent ongoing systemic infections
7. Illegal substance abuse, or social conditions that may interfere with patient's participation in the trial
8. Pre-existing neuropathy
9. Pregnant patients

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-12-12 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients eligible enrolled | 18 months
  Over an 18-month period The proportion of patients who complete the protocol (neoadjuvant therapy and pancreatectomy). As described, there are certain modifications of the neoadjuvant therapy protocol that are expected and allowed. The primary feasibility outcome will be one of the following:
  * Stop, main study non-feasible: 1) estimated proportion of eligible patients enrolled <40% or 2) estimated proportion of enrolled patients who complete the protocol (neoadjuvant therapy and pancreatectomy) <40%.
  * Continue with protocol modifications: 1) estimated proportion of eligible patients enrolled between 40-59% or 2) estimated proportion of enrolled patients who complete the protocol (neoadjuvant therapy and pancreatectomy) 40-59%.
  * Continue without modification: 1) estimated proportion of eligible patients enrolled equal to or greater than 60% or estimated proportion of enrolled patients who complete the protocol (neoadjuv

SECONDARY OUTCOMES:
Survival | 24 months
  Defined as percentage of patients alive at two years from enrolment.
Time to Progression | 24 months from the initiation of chemotherapy (the length of the study)
  Defined as the duration of time from enrolment to time to radiological evidence of disease progression or recurrence or death, whichever comes first.
Overall Complications from surgery | From date of surgery (POD=0) up to 90 postoperative days (POD=90)
  Occurrence of any postoperative complication (major or minor) from surgery following each patient's hospital stay and up to 90 days from the initial operation.
Pathological response to chemo-radiation treatment | From the date of the first chemotherapy to the date of surgery (around 4 months)
  Pathological response to treatment will be classified as per protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Leyo Ruo, MD, Principal Investigator — McMaster University
Locations (1):
- Juravinski Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No